CLINICAL TRIAL: NCT05007327
Title: Interaction Between Air Pollution, Pollens and Allergic Rhinitis in the Aix-Marseille-Provence Metropolis
Brief Title: Interaction Between Air Pollution, Pollens and Allergic Rhinitis
Acronym: MISTRAL
Status: Completed | Type: Observational
Sponsor: MASK-air SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: KM00111
Record Dates: First submitted 2021-05-19; First posted 2021-08-16 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2021-08

CONDITIONS: Allergic Rhinitis Due to Pollen; Allergic Rhinitis With Asthma
Keywords: Air pollution; Pollen; Allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — Air Pollution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exposure to pollen and air pollution — For all subjects of the cohort, we will follow exposure to pollen and air pollution.

SUMMARY:
Seasonal allergic rhinitis has multiple consequences: sleep disturbances, fatigue, depressed mood, impaired quality of life and productivity, and co-morbid conditions such as asthma, which affects one third of AR patients.

In Europe, more than 150 million people suffer from allergic rhinitis and more than 25 million suffer from asthma. About 30% have uncontrolled rhinitis during exposure to allergens. The impact of allergic diseases on work productivity is estimated to be between 30 and 50 billion € per year in the EU.

Studies show that pollution can play a role in the amplification of the response to inhaled pollen allergens by inducing morphological and functional modifications of nasal and bronchial epithelia, but also by inducing structural modifications of allergenic molecules. However, although data show that the symptoms of AR are aggravated by exposure to air pollution, this effect is not observed for all pollens.

The study area is very exposed to pollens (with a significant presence of cypress pollen) and air pollution, and presents a prevalence of asthma of 17% while the national average is about 7%.

The aim of this study is to establish, if they exist, links between pollens of various species, air pollution and symptoms of allergic rhinitis. The knowledge of these links will allow public authorities to set up prevention actions, and patients to better manage their allergic rhinitis on a daily basis.

DETAILED DESCRIPTION:
For this study, the investigators will collect real life data from volunteer citizens via the MASK-air® mobile application, and exposure data to air pollutants and pollens from their partners. The data will be collected over one year in order to cover all pollen seasons.

A communication of the project will be deployed to the citizens in the study area. The recruitment of participants will be done via an internet page accessible to all and presenting the MISTRAL study. Interested citizens can then access the electronic consent platform.

After signing the participation agreement, they will receive a link to download the MASK-air® mobile application (freely available via the Android and Apple stores) and a personal study code, which will allow them to install the application on their smartphone.

Participants will report their symptoms on the MASK-air app on a daily basis. Entry will only take 1 minute/day. This real-life data will be correlated with air pollution and pollen exposure data.

In anticipation of the prevention actions that will be deployed by the public authorities following this study, an analysis of the expectations and needs of the citizens will be carried out among a part of the participants in the form of 4 questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Person 18 years of age and older,
* Person suffering from seasonal allergic rhinitis (hay fever, pollen allergy),
* Person with an android and/or IOS smartphone and having the possibility to connect to the internet (via phone subscription or WIFI connection),
* Person agreeing to install the MASK-air application (medical device) on his personal smartphone,
* Person agreeing to activate their GPS when using the MASK-air® application for the study,
* Person having read and understood the information note and having signed their participation agreement prior to any specific study procedure.

Exclusion Criteria:

* Person who did not sign their participation agreement,
* Person who has difficulty understanding or reading the information note,
* Person planning to spend a significant percentage of time outside the area of interest (e.g., due to frequent business or personal travel),
* Person declaring to be under guardianship, curatorship or safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers living or spending significant time in the study area
Sampling Method: Non-Probability Sample
Enrollment: 1215 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in uncontrolled allergic rhinitis due to exposure to pollutants, exposure to pollens, and their interaction, as defined by VAS scores measuring the global discomfort and the use of medication in the MASK-air app. | Through the whole 1-year data collection period, an average participation of 30 days per participant is expected.
  A Visual Analogue Scale (VAS) measuring the global discomfort and the use of medication will be completed by the participants through the MASK-air mobile app.
  The minimum value of this VAS is 0 and means "no symptoms". The maximum value of the VAS is 100 and means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Charpin, Prof, Principal Investigator — Association pour la Prévention de la Pollution Atmosphérique
Locations (1):
- Https://Clin.Edop.Fr/Etude-Mistral, Montpellier, France

IPD SHARING:
Plan to Share IPD: No